CLINICAL TRIAL: NCT02133573
Title: Randomized Trial of Maternal Progesterone Therapy to Improve Neurodevelopmental Outcomes in Infants With Congenital Heart Disease
Brief Title: Randomized Trial of Maternal Progesterone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-010710
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Congenital Heart Disease; Periventricular Leucomalacia; Brain Development; Cardiac Surgery; Neurodevelopmental Disability; Fetal Neuroprotection
Keywords: progesterone; congenital heart disease; periventricular leucomalacia; brain development; cardiac surgery; neurodevelopmental disability; fetus; fetal neuroprotection
MeSH Terms: conditions — Heart Defects, Congenital; Leukomalacia, Periventricular | interventions — Progesterone; Replens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Experimental): Vaginal gel, 90mg twice a day (BID)
  Interventions: Drug: Progesterone
- Vaginal Lubricant (Placebo Comparator): Vaginal twice a day (BID)
  Interventions: Drug: Vaginal lubricant

INTERVENTIONS:
Drug: Progesterone — Crinone is supplied in a single use, disposable, white polypropylene vaginal applicator with a teal twist-off cap. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg (8% gel) of progesterone in a base containing glycerin, mineral oil, polycarbophil, carbomer 934P, hydrogenated palm oil glyceride, sorbic acid, purified water and may contain sodium hydroxide. Crinone 8% is administered vaginally at a dose of 90 mg twice daily. The rounded tip of the applicator is inserted into the vagina. After insertion, the plunger is pushed to release the gel into the vagina. The applicator is removed.
  Other Names: Crinone 8%
  Arms: Progesterone
Drug: Vaginal lubricant — Replens Long-Lasting Moisturizer is supplied in pre-filled, sealed and individually wrapped applicators.Replens Long-Lasting Moisturizer will also be dosed at one applicator intravaginally twice daily.
  Other Names: Replens
  Arms: Vaginal Lubricant

SUMMARY:
Neurodevelopmental disability is now recognized as the most common long-term complication after cardiac surgery in neonates. Research studies have shown that progesterone is critical to the development of the brain and in a variety of clinical situations including brain injury can protect the brain.

The purpose of this research study is to determine whether progesterone administered during the 3rd trimester of pregnancy (24-39 weeks) to pregnant women protects the brain of unborn babies with CHD and improves their neurodevelopmental outcomes after heart surgery.

DETAILED DESCRIPTION:
In the United States, approximately 1 in every 100 newborns is diagnosed with congenital heart disease (CHD). Many of these newborns (25%-35%) will require either corrective or palliative open heart surgery. As recently as the 1960's, only 20% of newborns with critical CHD survived to adulthood. Today, thanks to better diagnostic technologies and methods (including prenatal diagnosis), advances in surgery, and improved postoperative care, early survival is over 90%. However, with improved early outcomes has come the sobering recognition that there is an ongoing risk of late mortality, as well as significant morbidity for these children. In particular, neurodevelopmental disability is now recognized as the most common complication of critical CHD (i.e. those patients requiring cardiac surgery in infancy) and has the most negative impact on quality of life, academic performance and opportunity for independence as an adult.

The altered fetal hemodynamics secondary to CHD lead to decreased blood flow and/or oxygen delivery to the fetal brain. In turn, this impairment in blood flow and oxygenation results in impaired brain growth and altered structural and cellular maturation, particularly of the white matter. Fetal MRI studies have shown that during the third trimester, normally a time of rapid brain growth and development, brains of infants with CHD fail to grow at the same rate as the brains of fetuses without CHD. This growth delay results in microcephaly, immature cellular elements of the white matter and decreased cortical folding at birth. It has been demonstrated that brain immaturity at birth is a primary major risk factor underlying the hypoxic-ischemic white matter brain injury and subsequent neurodevelopmental disability seen in over 50% of infants following surgery for CHD. In addition, there is increasing evidence in the CHD population that even late pre-term birth (prior to 39 weeks GA) is associated with increased mortality, increased peri-operative morbidity, and worse neurodevelopmental outcomes.

Progesterone is an essential hormone in the occurrence and maintenance of pregnancy. Progesterone administration has also been shown to be neuroprotective in a variety of clinical situations, including traumatic brain injury (TBI). Sex steroid hormones, including progesterone, are critically involved in axonal myelination, forming the basis of white matter connectivity in the central nervous system (CNS). Progesterone and its metabolites not only promote the viability and regeneration of neurons, but also act on myelinating glial cell oligodendrocytes in the CNS and play an important role in the formation of myelin sheaths. Progesterone has also been shown to increase myelination and enhance maturation of immature oligodendrocytes progenitor cells to mature oligodendrocytes, which are more resistant to hypoxic/ischemic injury. Therapeutic administration of progesterone has also been demonstrated to prevent preterm birth. Thus, there are two potential mechanisms by which pre-natal progesterone therapy may improve neurodevelopmental outcomes in neonates with CHD: 1) a direct neuroprotective effect, and 2) decreasing the occurrence of pre-term birth.

Study Objectives

Primary: Develop preliminary evidence to support a multi-institutional study to determine whether, in women carrying fetuses (maternal-fetal dyad) with CHD, prophylactic vaginal natural progesterone therapy is neuroprotective, and compared to placebo improves neurodevelopmental outcomes at 18 months of age.

Secondary: Develop preliminary evidence to support a multi-institutional study to determine whether, in women carrying fetuses (maternal-fetal dyad) with CHD, prophylactic vaginal natural progesterone therapy is neuroprotective, and compared to placebo:

1. improves fetal brain growth and maturation,
2. increases myelination during fetal brain development,
3. reduces pre-operative brain white matter injury, and
4. reduces post-operative white matter injury.

ELIGIBILITY:
Inclusion Criteria: Mother carrying a fetus with CHD (maternal-fetal dyad) requiring surgery with cardiopulmonary bypass (CPB) prior to 44 weeks corrected gestational age (GA) identified prior to 28 weeks GA.

Exclusion Criteria:

1. Major genetic or extra-cardiac anomaly other than 22q11 deletion
2. Language other than English spoken in the home
3. Known sensitivity or listed contraindication to progesterone (known allergy or hypersensitivity to progesterone, severe hepatic dysfunction, undiagnosed vaginal bleeding, mammary or genital tract carcinoma, thrombophlebitis, thromboembolic disorders, cerebral hemorrhage, porphyria)
4. Prescription or ingestion of medications known to interact with progesterone (e.g. Bromocriptine, Rifamycin, Ketoconazole or Cyclosporin)
5. Maternal use of progesterone within 30 days of enrollment
6. History of preterm birth or short cervix (defined as cervical length ≤ 25 mm at 18-24 weeks GA necessitating progesterone therapy
7. Multiple gestation
8. Maternal contraindication for magnetic resonance imaging (MRI)
9. Subjects with a known history of non-compliance with medical therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-07; Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. William Gaynor, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gaynor JW, Moldenhauer JS, Zullo EE, Burnham NB, Gerdes M, Bernbaum JC, D'Agostino JA, Linn RL, Klepczynski B, Randazzo I, Gionet G, Choi GH, Karaj A, Russell WW, Zackai EH, Johnson MP, Gebb JS, Soni S, DeBari SE, Szwast AL, Ahrens-Nicklas RC, Drivas TG, Jacobwitz M, Licht DJ, Vossough A, Nicolson SC, Spray TL, Rychik J, Putt ME. Progesterone for Neurodevelopment in Fetuses With Congenital Heart Defects: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2412291. doi: 10.1001/jamanetworkopen.2024.12291. PMID 38805228
- See also: The Children's Hospital of Philadelphia Fetal Neuroprotection and Neuroplasticity Program — http://www.chop.edu/service/fetal-diagnosis-and-treatment/the-center-for-fetal-research/fetal-neuroprotection-neuroplasticity.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Cardiac Center at Children's Hospital of Philadelphia (CHOP) between July 2014 and February 2020.102 maternal subjects and their fetuses (dyads) were enrolled. On February 26, 2020 it was the unanimous opinion of the Data Safety Monitoring Board (DSMB) that enrollment in the trial should be stopped for futility.
Period: Overall Study
Arm/Group | Progesterone | Vaginal Lubricant
Started | 52 | 50
Dyads Allocated to Intervention | 52 | 49 (One participant had a maternal adverse event prior to initiating the allocated intervention.)
Number of Toddlers That Returned for 18 Month Follow Up Visit | 45 | 43
Number of Toddlers With Analyzed Primary Endpoint | 43 | 42
Completed | 43 | 42
Not Completed | 9 | 8
Not completed — Withdrawal by Maternal Subjects | 2 | 1
Not completed — Child Deaths | 3 | 5
Not completed — Child Declined Follow Ups | 2 | 1
Not completed — Child missing primary endpoint score due to child's inability to test | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants for each arm represent the number of dyads.
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Vaginal Lubricant | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age at the time of enrollment
  years | 30.35 (5.90) | 30.62 (4.40) | 30.48 (5.20)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age the progesterone or vaginal lubricant was initiated
  weeks | 27.8 (0.606) | 27.7 (0.597) | 27.8 (0.599)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 48 | 43 | 91
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 36 | 41 | 77
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 2 | 2
Marital Status [Count of Participants; unit: Participants]
  Single | 8 | 7 | 15
  Married | 43 | 43 | 86
  Divorced | 1 | 0 | 1
Mom Works Outside Home [Count of Participants; unit: Participants]
  Yes | 38 | 40 | 78
  No | 14 | 10 | 24
Income [Count of Participants; unit: Participants]
  Less than 25,000 | 3 | 1 | 4
  25,000-50,000 | 4 | 3 | 7
  51,000-75,000 | 5 | 7 | 12
  76,000-100,000 | 9 | 9 | 18
  Greater than 100,000 | 19 | 25 | 44
  Don't know | 5 | 2 | 7
  Prefer not to answer | 2 | 3 | 5
  Missing | 5 | 0 | 5
Maternal Education [Count of Participants; unit: Participants]
  Partial high school | 1 | 0 | 1
  Graduated high school (12th grade) | 6 | 3 | 9
  Partial college or trade school | 6 | 7 | 13
  College graduate | 17 | 26 | 43
  Post graduate degree | 22 | 14 | 36
Fetal Cardiac Diagnosis [Count of Participants; unit: Participants]
  Hypoplastic Left Heart Syndrome (HLHS) | 27 | 25 | 52
  Transposition of the Great Arteries (TGA) | 19 | 19 | 38
  OTHER | 6 | 6 | 12
Child Genetic Classification [Count of Participants; unit: Participants]
  Normal | 29 | 32 | 61
  Suspect | 12 | 5 | 17
  Abnormal | 9 | 11 | 20
  Unknown | 0 | 1 | 1
  Missing | 2 | 1 | 3
Child 22q11.2 Deletion [Count of Participants; unit: Participants]
  Yes | 4 | 1 | 5
  No | 46 | 47 | 93
  Unknown | 0 | 1 | 1
  Missing | 2 | 1 | 3
Child Apolipoprotein E (APOE) Haplotype [Count of Participants; unit: Participants]
  E2 | 8 | 6 | 14
  E2/E4 | 0 | 1 | 1
  E3 | 26 | 30 | 56
  E4 | 14 | 10 | 24
  Missing | 4 | 3 | 7
Paternal Race [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Black/African American | 5 | 6 | 11
  White | 38 | 41 | 79
  Not known | 0 | 1 | 1
  Choose not to answer | 0 | 1 | 1
  Missing | 3 | 1 | 4
  Multiple | 3 | 0 | 3
Paternal Hispanic Ethnicity [Count of Participants; unit: Participants]
  Yes | 1 | 6 | 7
  No | 47 | 42 | 89
  Choose not to answer | 0 | 2 | 2
  Missing | 4 | 0 | 4
Dad Employed [Count of Participants; unit: Participants]
  Yes | 50 | 47 | 97
  No | 1 | 2 | 3
  Missing | 1 | 1 | 2
Paternal Education [Count of Participants; unit: Participants]
  Graduated high school (12th grade) | 10 | 8 | 18
  Partial college or trade school | 9 | 13 | 22
  College graduate | 18 | 18 | 36
  Post graduate degree | 12 | 10 | 22
  Refused to answer | 1 | 0 | 1
  Missing | 2 | 1 | 3
Child Race [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Black/African American | 6 | 3 | 9
  White | 34 | 40 | 74
  Choose not to answer | 0 | 1 | 1
  Missing | 2 | 1 | 3
  Multiple | 7 | 5 | 12
Child Hispanic Ethnicity [Count of Participants; unit: Participants]
  Yes | 2 | 7 | 9
  No | 47 | 41 | 88
  Choose not to answer | 0 | 1 | 1
  Missing | 3 | 1 | 4
Child Gender [Count of Participants; unit: Participants]
  Male | 34 | 31 | 65
  Female | 16 | 18 | 34
  Missing | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Motor Scale of the Bayley Scales of Infant and Toddler Development-III
Description: The composite motor score is normed and has a mean of 100 (SD 15) and a range of 40-160. Scores between 71 and 85 indicate mild impairment and scores lower than 70 indicate moderate or severe impairment.
Time Frame: When baby is 18 months of age
Population: Per protocol population, all children who completed the 18 month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overall: Treatment 1 and Treatment 2 Combined
Arm/Group | Progesterone | Vaginal Lubricant | Overall
Number analyzed (Participants) | 45 | 43 | 88
score on a scale | 90.0 (11.5) | 87.5 (12.7) | 88.7 (12.1)

2. Secondary Outcome: Cognitive and Language Scales of the Bayley Scale of Infant and Toddler Development-III
Description: The composite cognitive and language scores are normed and have a mean of 100 (SD 15) and a range of 40-160. Scores between 71 and 85 indicate mild impairment and scores lower than 70 indicate moderate or severe impairment.
Time Frame: When baby is 18 months of age
Population: Per protocol population, all children who completed the 18 month follow up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Overall: Progesterone and Vaginal Lubricant Arms Combined
Arm/Group | Progesterone | Vaginal Lubricant | Overall
Number analyzed (Participants) | 45 | 43 | 88
score on a scale
  Bayley Cognitive Score (Composite) | 92.4 (12.2) | 91.2 (11.4) | 91.8 (11.8)
  Bayley Language Score (Composite) | 86.1 (15.1) | 84.5 (18.9) | 85.3 (16.9)

3. Secondary Outcome: Fetal Brain Growth and Maturation by MRI
Description: Total maturation scale (TMS) is an observational rating scale to assess the appropriateness of the gross brain appearance on MRI. The TMS scale has been used to demonstrate the negative effect of heart anatomy on post-natal, pre-surgical brain MRIs in infants with congenital heart. Similarly, a fetal TMS scale (fTMS) was developed to define the progress of brain development in-utero. Here we use the fTMS to define developmental/maturational changes occurring during gestation. The fTMS was graded on an ordinal scale, minimum = 4, maximum = 17 where a lower number indicates a less mature fetal brain and a higher number indicates a more mature fetal brain on MRI.
Time Frame: fTMS score change from 24-28 weeks gestational age to 34-36 weeks gestational age
Population: Number of participants who completed both fetal MRIs and had reliable TMS scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progesterone | Vaginal Lubricant
Number analyzed (Participants) | 31 | 29
score on a scale | 8.84 (1.19) | 8.35 (1.27)

4. Secondary Outcome: Myelination During Fetal Brain Development by MRI
Description: Myelination is part of the fetal TMS rating system and is scored as follows.
  1. - If there is myelin in the brainstem, cerebellar peduncle and inferior tectum only
  2. - If there is myelin in the ventrolateral thalamus as well as in #1
  3. - If there is myelin present in the posterior limb of the internal capsule as well as in #2
Time Frame: Change from 24-28 weeks gestational age to 34-36 weeks gestational age
Population: Number of participants who completed both fetal MRIs and had reliable myelination scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Progesterone | Vaginal Lubricant
Number analyzed (Participants) | 32 | 29
score on a scale | 0.72 (0.5) | 0.69 (0.4)

5. Secondary Outcome: Prevalence of PVL/WMI in the Pre Operative Study Participants
Description: Periventricular leukomalacia (PVL), also known in the literature as white matter injury (WMI), is an acquired brain injury to the white matter of the brain seen in 20% of infants with congenital heart and up to 80% post-operatively. PVL/WMI is seen on T1 MPR sequences as abnormal hyperintensities in the white matter which are quantified by manual segmentation to achieve total volumes and regional volumes of the injury. Yes indicates the presence of PVL and no indicates the absence of PVL on the pre operative MRI.
Time Frame: Preoperative on day of surgery
Population: The number of participants who completed a pre operative MRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Vaginal Lubricant | Overall
Number analyzed (Participants) | 35 | 34 | 69
Participants
  Yes | 8 | 9 | 17
  No | 27 | 25 | 52

6. Secondary Outcome: Prevalence of PVL/WMI in the Post Operative Study Participants
Description: PVL/WMI will be measured on the post operative brain MRI with manual segmentations from the T1MPR sequence. Yes indicates the presence of new or worse PVL and no indicates the absence of new or worse PVL on the post operative MRI.
Time Frame: Postoperative within 10 days of surgery
Population: The number of participants who completed a post operative MRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Progesterone | Vaginal Lubricant | Overall
Number analyzed (Participants) | 37 | 36 | 73
Participants
  Yes | 18 | 15 | 33
  No | 19 | 21 | 40

ADVERSE EVENTS:
Time Frame: Maternal adverse event data was collected from randomization through delivery, an average of 12 weeks. Child adverse event data was collected from birth through their follow up visit, an average of 18 months.
Description: Maternal adverse events were collected using Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v.4.0)
  Child adverse events were collected using Pediatric Heart Network: Single Ventricle Reconstruction Trial Code List M: Complications and Sentinel Serious Events Version A (PHN Code List M)
  All adverse event terms corresponding to the mothers and the children are reported separately, even if they repeat, as indicated by the associated source vocabulary name for each term.
Groups:
- Progesterone (Maternal Adverse Events); Progesterone (Child Adverse Events): Vaginal gel, 90mg twice a day (BID)
  Progesterone: Crinone is supplied in a single use, disposable, white polypropylene vaginal applicator with a teal twist-off cap. Each applicator delivers 1.125 grams of Crinone gel containing 90 mg (8% gel) of progesterone in a base containing glycerin, mineral oil, polycarbophil, carbomer 934P, hydrogenated palm oil glyceride, sorbic acid, purified water and may contain sodium hydroxide. Crinone 8% is administered vaginally at a dose of 90 mg twice daily. The rounded tip of the applicator is inserted into the vagina. After insertion, the plunger is pushed to release the gel into the vagina. The applicator is removed.
- Vaginal Lubricant (Maternal Adverse Events); Vaginal Lubricant (Child Adverse Events): Vaginal twice a day (BID)
  Vaginal lubricant: Replens Long-Lasting Moisturizer is supplied in pre-filled, sealed and individually wrapped applicators.Replens Long-Lasting Moisturizer will also be dosed at one applicator intravaginally twice daily.
Arm/Group | Progesterone (Maternal Adverse Events) | Vaginal Lubricant (Maternal Adverse Events) | Progesterone (Child Adverse Events) | Vaginal Lubricant (Child Adverse Events)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 3/50 | 5/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/50 | 46/50 | 43/49
Other Adverse Events (participants affected / at risk) | 51/52 | 48/50 | 48/50 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Progesterone (Maternal Adverse Events) (N=52) | Vaginal Lubricant (Maternal Adverse Events) (N=50) | Progesterone (Child Adverse Events) (N=50) | Vaginal Lubricant (Child Adverse Events) (N=49)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Uterine Hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Uterine Atony (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Listing for Cardiac Transplant (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
Thromboelic Event (Vascular disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
Heart Block (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
Need for Surgical or Catheter-Based Intervention (Surgical and medical procedures) | 0/0 (0) | 0/0 (0) | 46 (131) | 41 (115)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Progesterone (Maternal Adverse Events) (N=52) | Vaginal Lubricant (Maternal Adverse Events) (N=50) | Progesterone (Child Adverse Events) (N=50) | Vaginal Lubricant (Child Adverse Events) (N=49)
Vaginal Discharge (Reproductive system and breast disorders) | 33 (43) | 32 (38) | 0/0 (0) | 0/0 (0)
Uterine Pain (Reproductive system and breast disorders) | 11 (14) | 12 (13) | 0/0 (0) | 0/0 (0)
Vaginal Pain (Reproductive system and breast disorders) | 12 (12) | 14 (15) | 0/0 (0) | 0/0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 9 (9) | 0/0 (0) | 0/0 (0)
Headache (Nervous system disorders) | 10 (12) | 7 (7) | 0/0 (0) | 0/0 (0)
Vaginal Infection (Infections and infestations) | 9 (11) | 6 (6) | 0/0 (0) | 0/0 (0)
Hypertension (Vascular disorders) | 10 (10) | 7 (7) | 0/0 (0) | 0/0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 8 (8) | 7 (7) | 0/0 (0) | 0/0 (0)
Edema Limbs (General disorders) | 5 (6) | 6 (6) | 0/0 (0) | 0/0 (0)
Fatigue (General disorders) | 8 (8) | 4 (4) | 0/0 (0) | 0/0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8) | 0/0 (0) | 0/0 (0)
Premature Delivery (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 6 (6) | 0/0 (0) | 0/0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 4 (4) | 0/0 (0) | 0/0 (0)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 5 (5) | 5 (5) | 0/0 (0) | 0/0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 0/0 (0) | 0/0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3) | 0/0 (0) | 0/0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 0/0 (0) | 0/0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (6) | 2 (2) | 0/0 (0) | 0/0 (0)
Uterine Hemorrhage (Reproductive system and breast disorders) | 4 (4) | 4 (4) | 0/0 (0) | 0/0 (0)
Vaginal Inflammation (Reproductive system and breast disorders) | 6 (7) | 1 (1) | 0/0 (0) | 0/0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0/0 (0) | 0/0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0/0 (0) | 0/0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (4) | 2 (2) | 0/0 (0) | 0/0 (0)
Psychiatric Disorders - Other (Psychiatric disorders) | 3 (3) | 3 (3) | 0/0 (0) | 0/0 (0)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 5 (5) | 0/0 (0) | 0/0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 3 (3) | 0/0 (0) | 0/0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 0/0 (0) | 0/0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0/0 (0) | 0/0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0/0 (0) | 0/0 (0)
Skin and Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0/0 (0) | 0/0 (0)
Blurred Vision (Eye disorders) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Fetal Growth Retardation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Libido Increased (Psychiatric disorders) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Breast Pain (Reproductive system and breast disorders) | 2 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0/0 (0) | 0/0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0/0 (0) | 0/0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0/0 (0) | 0/0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Breast Infection (Infections and infestations) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0/0 (0) | 0/0 (0)
Reproductive System and Breast Disorders - Other (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0/0 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0/0 (0) | 0/0 (0)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Flashing Lights (Eye disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Flu Like Symptoms (General disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Conjunctivitis Infective (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Infections and Infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Intraoperative Reproductive Tract Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Metabolism and Nutrition Disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Nervous System Disorders - Other (Nervous system disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Bladder Spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Renal Calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Renal and Urinary Disorders - Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Lactation Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Respiratory, Thoracic and Mediastinal Disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Surgical and Medical Procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
Hot Flashes (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Superficial Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0/0 (0) | 0/0 (0)
Vascular Disorders - Other (Vascular disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0/0 (0)
M-0001 Atrial fibrillation (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
M-0002 Atrial Flutter (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
M-0003 Supraventricular Tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 13 (16) | 8 (8)
M-0004 Junctional Ectopic Tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 3 (3)
M-0005 Sinus node dysfunction (requiring pacing) (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 4 (6) | 3 (3)
M-0006 Atrioventricular block (second or third, not first) (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 0 (0)
M-0007 Ventricular tachycardia (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 2 (3)
M-0008 Ventricular fibrillation (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 3 (4)
M-0020 Hemopericardium (requiring intervention) (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
M-0021 Pericardial effusion (requiring drainage) (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
M-0030 Hypotension (<40mmHg for neonates; <50 mmHg after Stage II) (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 9 (12) | 11 (14)
M-0099 Other Cardiac (Cardiac disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 5 (7)
M-0101 Chronic respiratory failure (intubated for >2 weeks after surgery) (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 4 (4)
M-0102 Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 7 (10) | 4 (5)
M-0103 Diaphragm paralysis (fluoro or ultrasound) (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 2 (2)
M-0104 Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
M-0105 Phrenic nerve injury (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
M-0106 Pleural effusion requiring drainage (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 11 (16) | 5 (5)
M-0107 Pneumothorax requiring tube insertion (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 1 (1)
M-0109 Vocal cord injury (direct visualization) (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 7 (7) | 2 (2)
M-0199 Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
M-0201 Abnormal head CT scan (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 7 (11) | 1 (1)
M-0202 Abnormal head MRI scan (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 35 (49) | 35 (53)
M-0205 Intracranial bleeding (confirmed by imaging) (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 32 (41) | 33 (36)
M-0206 Seizure(s) - definite (EEG or obvious motor) (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 9 (12) | 7 (7)
M-0207 Stroke (confirmed by imaging study) (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 11 (11) | 3 (3)
M-0299 Other, Neurological (Nervous system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (1)
M-0301 Cholestasis (Direct bilirubin >4) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 2 (2)
M-0302 Hyperbilirubinemia (requiring phototherapy or direct bilirubin >5) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 4 (4)
M-0303 Liver failure (AST, ALT or GGT >500) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 4 (4) | 3 (4)
M-0304 NEC, confirmed (pneumatosis or free air) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 3 (3)
M-0305 NEC, suspected (NPO, antibiotics started) (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 3 (4)
M-0399 Other, Gastrointestinal (Gastrointestinal disorders) | 0/0 (0) | 0/0 (0) | 20 (22) | 16 (17)
M-0403 Line Infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (1)
M-0404 Mediastinitis (Infections and infestations) | 0/0 (0) | 0/0 (0) | 2 (2) | 1 (1)
M-0405 Sepsis, confirmed (positive blood culture, not line infection) (Infections and infestations) | 0/0 (0) | 0/0 (0) | 3 (4) | 3 (3)
M-0406 Sepsis, suspected (antibiotics started) (Infections and infestations) | 0/0 (0) | 0/0 (0) | 25 (47) | 24 (43)
M-0407 Wound infection, superficial (Infections and infestations) | 0/0 (0) | 0/0 (0) | 10 (10) | 10 (10)
M-0499 Other infection (Infections and infestations) | 0/0 (0) | 0/0 (0) | 7 (7) | 7 (9)
M-0501 Acute renal failure (creatinine >1.5 or tripling of baseline value for <7 days) (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 4 (4)
M-0502 Chronic renal failure (creatinine >1.5 or tripling of baseline value for >7 days) (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (2)
M-0503 Hemodialysis (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 2 (2)
M-0504 Peritoneal dialysis (Renal and urinary disorders) | 0/0 (0) | 0/0 (0) | 0 (0) | 1 (2)
M-0601 Anemia (Hemoglobin <10 gm/dl) (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 19 (33) | 17 (25)
M-0602 Thrombocytopenia (plts <50,000) (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 11 (16) | 9 (16)
M-0603 Thrombus/thromboembolism (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 11 (14) | 11 (20)
M-0699 Other, Hematologic (Blood and lymphatic system disorders) | 0/0 (0) | 0/0 (0) | 1 (1) | 1 (2)
M-9999 Other, Misc (General disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02133573/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT02133573/SAP_001.pdf